CLINICAL TRIAL: NCT01924455
Title: HBV-HIV Coinfection Research Network
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20000444; DK094818 (Other: NIH)
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis B; Human Immunodeficiency Virus
Keywords: HIV; HBV
MeSH Terms: conditions — Hepatitis B; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum at baseline and every 6 months for 4 years. Liver biopsy at baseline and year 4
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HBV-HIV coinfected subjects: HBV-HIV coinfected subjects seen at one of 7 participating centers.

SUMMARY:
Despite effective ART that can suppress both HIV and HBV, HBV-related liver disease remains a significant co-morbidity in this population. Little is known about the histologic spectrum of liver disease, the significance of complete vs. incomplete HBV suppression, the utility of novel virologic and serum markers of disease severity, and the long-term renal and bone effects of TDF-based therapy. This proposal will address these important questions and impact the science and health of those coinfected with HBV-HIV.

DETAILED DESCRIPTION:
Since the introduction of highly active antiretroviral therapy (ART) in 1996, there has been a dramatic reduction in morbidity and mortality among those living with HIV. However, chronic liver disease due to coinfection with hepatitis B (HBV) or C (HCV) virus has emerged as the second leading cause of mortality among HIV-infected persons. The natural history of HBV infection is altered in those with HIV. Current guidelines recommend that most coinfected patients be treated for both HIV and HBV infection using combinations of ART that include tenofovir (TDF). Despite widespread adoption in the US, the effect of this regimen on long-term outcomes of HBV disease such as histologic severity, progression, and risk of emergence of resistant HBV variants, and the long term risks of TDF therapy remains unanswered. Further investigation is required to address the following important questions: (1) what is the proportion of HIV-coinfected patients who have incomplete viral suppression on TDF?; (2) is incomplete suppression of HBV acceptable in HIV coinfected persons and if so, what threshold HBV DNA level constitutes an adequate clinical goal?; (3) in view of the lack of acceptance of liver biopsy among HIV practitioners, can noninvasive markers accurately assess HBV disease activity and the impact of ART on disease progression?; (4) What are the long term risks of TDF-based therapy for HBV in HIV coinfection? In short, what are the risks and benefits of TDF-based therapy for CHB in patients with HIV coinfection? The NIH Hepatitis B Research Network (HBRN) is the first major effort to elucidate the natural history and treatment outcomes of persons with chronic HBV the US. The HBRN will not address the critical issue of HBV liver disease progression in HIV-infected persons because patients with HIV coinfection will be excluded. The current proposal, an approved ancillary study of the HBRN, offers a unique opportunity to fill major gaps in HBV-HIV knowledge and to compare HBV-HIV infected persons to those with HBV monoinfection participating in the HBRN. No other funded research network in North America has the expertise, patient population, and structure to carry out the proposed studies. The Specific Aims are: 1. Define the problem. We will clinically, histologically, serologically, and virologically characterize a well-defined cohort of HBV-HIV patients in North America in a cross-sectional manner; 2. Define the benefit of long term therapy. We will longitudinally determine the impact of complete vs. incomplete viral suppression on clinical and serologic outcomes, and histologic progression by paired biopsy and 2a. Define a threshold HBV DNA level associated with disease progression; 2b. Establish the utility of noninvasive assessment of hepatic fibrosis compared with biopsy; and 2c. Define the frequency of genotypic and phenotypic TDF resistance with long term therapy; and finally 3. Define the risk of long term therapy. We will assess the long term renal and bone effects of TDF-based therapy in the HBV-HIV cohort. Collectively, this study will fulfill many of the key priorities outlined in the NIH Action Plan for Liver Disease for HBV-HIV coinfection.

ELIGIBILITY:
Inclusion Criteria: (1) Male and female subjects ≥ 18 years of age; (2) Serologic evidence of HIV infection by HIV antibody positivity or positive HIV-RNA > 6 months prior to screening (3) Serologic evidence of chronic hepatitis B infection by HBsAg positivity(4) Willingness to provide informed consent.

-

Exclusion Criteria: (1) Estimated life expectancy of less than one year based on clinical judgment of the investigator; (2) Hepatic decompensation as defined by presence of ascites or hepatic hydrothorax, variceal or portal hypertensive bleeding, hepatic encephalopathy, or Child-Turcotte-Pugh (CTP) score of 7 or above; (3) Hepatocellular carcinoma (HCC); (4) Anti-HCV positive; (5) History of solid organ or bone marrow transplantation; (6) Pregnant women; (7) Medical or social condition which in the opinion of the study physician would make the patient unsuitable for the study or will interfere with or prevent follow-up per protocol; (8) Unable or unwilling to return for follow-up visits; (9) Contraindications to liver biopsy.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV-HIV coinfection
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-04; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Liver disease severity | 4 years
  We will clinically, histologically, serologically, and virologically characterize a well-defined cohort of HBV-HIV patients in North America in a cross-sectional manner

SECONDARY OUTCOMES:
Outcome of viral suppression | 4 years
  1. We will longitudinally determine the impact of complete vs. incomplete viral suppression on clinical and serologic outcomes, and histologic progression by paired biopsy.
  2. Define a threshold HBV DNA level associated with disease progression.
  3. Establish the utility of noninvasive assessment of hepatic fibrosis compared with biopsy.
  4. Define the frequency of genotypic and phenotypic TDF resistance with long term therapy
  5. We will assess the long term renal and bone effects of TDF-based therapy in the HBV-HIV cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sterling, MD, MSc, Principal Investigator — Virginia Commonwealth University
Locations (8):
- United States (7):
  - University of California, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - NIDDK, Bethesda, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - UT Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Toronto Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lisker-Melman M, King WC, Ghany MG, Chung RT, Hinerman AS, Cloherty GA, Khalili M, Jain MK, Sulkowski M, Sterling RK. Human immunodeficiency virus coinfection differentially impacts hepatitis B virus viral markers based on hepatitis Be antigen status in patients with suppressed viremia. J Viral Hepat. 2023 Aug;30(8):700-709. doi: 10.1111/jvh.13857. Epub 2023 Jun 6. PMID 37278302
- [Derived] Lisker-Melman M, Wahed AS, Ghany MG, Chung RT, King WC, Kleiner DE, Bhan AK, Khalili M, Jain MK, Sulkowski M, Wong DK, Cloherty G, Sterling RK. HBV transcription and translation persist despite viral suppression in HBV-HIV co-infected patients on antiretroviral therapy. Hepatology. 2023 Feb 1;77(2):594-605. doi: 10.1002/hep.32634. Epub 2022 Jul 21. PMID 35770681
- [Derived] Sterling RK, King WC, Khalili M, Chung RT, Sulkowski M, Jain MK, Lisker-Melman M, Ghany MG, Wong DK, Hinerman AS, Bhan AK, Wahed AS, Kleiner DE; HBV-HIV Cohort Study of the Hepatitis B Research Network. A Prospective Study Evaluating Changes in Histology, Clinical and Virologic Outcomes in HBV-HIV Co-infected Adults in North America. Hepatology. 2021 Sep;74(3):1174-1189. doi: 10.1002/hep.31823. Epub 2021 Aug 25. PMID 33743541
- [Derived] Sterling RK, King WC, Khalili M, Kleiner DE, Hinerman AS, Sulkowski M, Chung RT, Jain MK, Lisker-Melman MA, Wong DK, Ghany MG; HBV-HIV Cohort Study of the Hepatitis B Research Network. Performance of Serum-Based Scores for Identification of Mild Hepatic Steatosis in HBV Mono-infected and HBV-HIV Co-infected Adults. Dig Dis Sci. 2022 Feb;67(2):676-688. doi: 10.1007/s10620-021-06860-3. Epub 2021 Feb 8. PMID 33559089
- [Derived] Khalili M, King WC, Kleiner DE, Jain MK, Chung RT, Sulkowski M, Lisker-Melman M, Wong DK, Ghany M, Sanyal A, Sterling RK. Fatty Liver Disease in a Prospective North American Cohort of Adults With Human Immunodeficiency Virus and Hepatitis B Virus Coinfection. Clin Infect Dis. 2021 Nov 2;73(9):e3275-e3285. doi: 10.1093/cid/ciaa1303. PMID 32869840
- [Derived] Sterling RK, King WC, Wahed AS, Kleiner DE, Khalili M, Sulkowski M, Chung RT, Jain MK, Lisker-Melman M, Wong DK, Ghany MG; HIV-HBV Cohort Study of the Hepatitis B Research Network. Evaluating Noninvasive Markers to Identify Advanced Fibrosis by Liver Biopsy in HBV/HIV Co-infected Adults. Hepatology. 2020 Feb;71(2):411-421. doi: 10.1002/hep.30825. Epub 2019 Aug 19. PMID 31220357
- See also: HBRN website — http://www.hepbnet.org/

DOCUMENTS (1):
  • Informed Consent Form (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT01924455/ICF_000.pdf